CLINICAL TRIAL: NCT05458557
Title: Evaluation of Antigen Rapid Diagnostic Tests (Ag-RDTs) for Community Identification of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) in Kiambu County, Kenya
Brief Title: Antigen Rapid Diagnostic Tests for Community Identification of Severe Acute Respiratory Syndrome Coronavirus 2
Status: Completed | Type: Observational
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Find (Other); Kiambu County (Unknown)
Responsible Party: Principal Investigator, Rose Otieno Masaba, Associate Director Public Health Evaluations, Elizabeth Glaser Pediatric AIDS Foundation
Other Study IDs: EG0278
Record Dates: First submitted 2022-07-07; First posted 2022-07-14 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — naso-pharyngial swabs collected for purposes of identification of SARS-COV-2
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rapid Antigen Testing — Community testing for SARS-COV-2 using rapid Antigen test

SUMMARY:
Background:

Background: Testing with antigen-detecting rapid diagnostic tests (Ag-RDTs), including in asymptomatic individuals, has the potential to promptly identify more Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infections and consequently decrease spread of coronavirus-19 disease at the community level. In addition, rapid test results are important for immediate clinical management and isolation of patients with SARS-CoV-2 infection, and for contact tracing and quarantining of contacts. Data on SARS-CoV-2 infection rates, the acceptability of Ag-RDT, and the cost of conducting widespread testing in these communities are limited in Africa.

Study Aim and Objectives: To generate evidence evaluating the use of Ag-RDTs for community identification of SARS-CoV-2 infections within large gathering venues such as work places, schools, places of worship, and markets.

The primary objective is to determine the SARS-CoV-2 case detection rate through a mass testing approach in large gatherings. Secondary objectives include determining the proportion of asymptomatic and symptomatic infections detected, acceptance of mass SARS-CoV-2 Ag-RDT testing, the prevalence of circulating variants, and the cost of implementing this community testing strategy.

Study Design: The investigators propose a serial cross-sectional study design targeting approximately 15,000 persons, who will be offered testing in up to 50 different high attendance venues of Kiambu County that will be identified as possible points of community-based transmission. The study will follow an opt-in consent approach, with those accepting to participate providing additional information to the trained research assistant and/or health worker.

Outcome: Evidence will be generated to provide recommendations to the Kenya Ministry of Health, and more broadly to inform the field on the use of Ag-RDTs for large scale community screening by identifying best practices and stratifying risk areas for community transmission based on rates of infections detected within various settings.

DETAILED DESCRIPTION:
Study context

Since 31 March 2020, when the first case was confirmed in the country, a total of 20144 confirmed cases and 877 deaths (case fatality rate of (4.4%) have been line-listed as of 27th February 2022. Kiambu ranks second in cumulative number of confirmed Coronavirus-19 cases. Kiambu county has major gaps in Coronavirus-19 management due to inadequate resources limiting response capacity in detecting, investigating, contact tracing and follow up both in the facilities and within the community. The county has reported spikes in cases of Coronavirus-19 following participation in mass gathering events like in political rallies, markets, churches, burials, etc. The county has several tertiary institutions which have also been identified as high transmission hotspots. Kiambu county implements the Coronavirus-19 guidelines as stipulated in the ministry of health guidelines (hand washing, social distancing, use of masks etc), but non-compliance with Coronavirus-19 protocols has been noted in learning institutions and public places like Bus parks, markets and supermarkets.

The Elizabeth Glaser Pediatric AIDS Foundation (EGPAF) is supporting the Ministry of Health (MOH) in Kenya to accelerate an effective Coronavirus-19 response through novel solutions to increase access to high quality diagnostics and therapeutics through the Unitaid-funded Catalysing Coronavirus-19 Action (CCA) project. As part of this project, EGPAF is supporting decentralizing testing through integration of severe acute respiratory syndrome Coronavirus-2 (SARS-CoV-2) antigen rapid diagnostic test (Ag RDT) into Maternal Newborn Child Health, Tuberculosis and HIV clinics in about 31 facilities of Kiambu county. The project also enhances linkage to care and treatment including new therapeutics through a hub and spoke model. EGPAF works with civil society organizations and other key stakeholders in Kiambu county to increase demand for SARS-CoV-2 testing and care and treatment. This study will build upon the programmatic components of the CCA project to explore the effectiveness of SARS-CoV-2 AgRDT mass testing in high volume community venues to detect SARS-CoV-2 infections. The CCA project has been implemented since October 2021 with testing using Ag-RDT since January 2022 in Kiambu county. It has been observed that a number of clients attending facilities in services where the test is not currently offered are asking for testing, and during community vaccination campaigns, people are asking for the possibility to be tested.

Study Rationale As of 14 March 2022, 28.8% of adults were fully vaccinated in Kenya 4. Until vaccines have widespread availability, testing and isolation are the best methods to control disease spread at the national level. The use of simple, rapid, and affordable Ag-RDT to expand access to SARS-CoV-2 testing is being incorporated in many national Coronavirus-19 responses. Targeting high volume community venues has the potential to screen a lot of people within a limited amount of time and determine areas that are contributing to community transmission. Data on acceptability of mass SARS-CoV-2 Ag-RDT testing in these community settings in Africa are limited.

Most current programs use a screen and test strategy to identify symptomatic infection and those at risk due to exposure because of the limited availability and costs of broader testing. However, this strategy does not identify those with asymptomatic infection who also contribute to the spread of SARS-CoV-2 infection. Data are needed to inform the evolving SARS-CoV-2 testing guidelines and provide MOH with feasible and costed testing models to address their national strategies. This study will generate the evidence needed to determine the SARS-CoV-2 case detection rate and proportion of asymptomatic and symptomatic infections detected in high volume community venues using SARS-CoV-2 Ag-RDTs. Additionally, full genome sequencing of positive cases will be useful to the MoH in determining the circulating genomic strains in Kenya at real time and may contribute to national guidance.

Study Aim:

The aim of this study is to generate evidence evaluating the use of Ag-RDTs for community identification of SARS-CoV-2 infections within large gathering venues, and ultimately to determine if mass testing in such venues is a feasible and useful approach.

Primary Objective:

1.To estimate the SARS-CoV-2 case detection rate (number of SARS-CoV-2 infections detected per 100 individuals tested) in high volume community venues using SARS-CoV-2 Ag-RDT, overall and disaggregated by venue type.

Secondary Objectives:

To determine the number and proportion of venue attendees across the SARS-CoV-2 testing cascade: people offered Ag-RDT, who accept testing, receive test results, test positive, To determine the number and proportion of people who test positive with SARS-CoV2 RDT who are symptomatic, are referred for polymerase chain reaction (PCR) testing and confirmed with PCR, are referred for home-based isolation or care, To identify factors that are associated with SARS-CoV-2 infection, such as age, venue, exposure history and vaccination status.

To describe SARS-CoV-2 variants among SARS-CoV-2 positive attendees To determine costs associated with implementation of SARS-CoV-2 Ag-RDT in community settings.

The investigators hypothesize that with the introduction of SARS-CoV-2 mass testing in high-exposure venues in the community, more individuals will have access to testing services, individuals will accept SARS-CoV-2 Ag RDT, symptomatic and asymptomatic SARS-CoV-2 infections will be diagnosed, and individuals diagnosed with SARS-CoV-2 will be linked to care and treatment services. This will lead to isolation of SARS-CoV-2 infected individuals, quarantining of contacts, and medical treatment for those requiring it.

Study Design This will be a community-based cross-sectional study. The study will be conducted among the population of Kiambu County, central Kenya, attending specific high-volume community venues identified as possible points of community-based transmission.

These high-volume community venues will be:

Venues identified by individuals diagnosed with SARS-CoV-2 infection in a subset of CCA-supported facilities in Kiambu County. As part of the CCA questionnaire, participants will be asked to identify crowded places the participants had been to in the 10 days prior to their positive SARS-CoV-2 test. This will provide an opportunity for the staff to identify market places, places of worship, schools, or other venues where SARS-CoV-2 transmission is likely to occur in the communities. In this study, no testing activities will be conducted in health facilities.

Venues identified in collaboration with the department of public health and the Coronavirus-19 response team in the county that may act as transmission hotspots.

Using both approaches above, the investigators will identify venues in Kiambu county where a large number of people congregate to propose mass testing.

Variant surveillance population Individuals who test positive with SARS-Cov-2 Ag-RDT and those who test negative but with symptoms of Coronavirus-19 will be asked to provide a second sample for confirmatory PCR testing and whole genome sequencing for variant surveillance. The participants will be taken care of as Coronavirus-19 cases as the participant wait for the PCR result. Based on the national guidelines on management of Coronavirus-19 in Kenya, a person who meets the clinical and epidemiological criteria is a suspected case of SARS-CoV-2. The participant will be assessed and based on the severity of their symptoms the participant will either be referred to a treatment centre where symptoms will be managed. If the person has mild symptoms he will be referred for home based care. The study team will transport those who need to be hospitalized to the hospital. Kiambu county currently has 5 treatment centres which also act as isolation centres. While secondary sample collection is part of routine national surveillance, because these results will be used for research purposes, the investigators will only perform this study activity for those who voluntarily agree to this study through administration of a written informed consent. The second sample will be taken at the community venue for those who will have given written consent/assent and transported to the testing laboratory in accordance with the standard operating procedures.

Inclusion criteria for variant surveillance:

Venue attendee with a positive result to SARS-Cov-2 Ag-RDT Venue attendee with a negative Ag-RDT, but with Coronavirus-19 symptoms Provide written informed consent to collect a second sample Community mobilization and recruitment This section describes activities conducted by Kiambu County Coronavirus-19 response team ahead of the start of study activities.

Mobilizing the community to ensure a high response rate is a priority for successful study implementation the Kiambu County Coronavirus-19 response team will be engaged from the initial stages to ensure that the security coordination mechanisms are well informed.

Before the mass testing, meetings will be held with the community leaders to explain the study and have the opportunity to discuss potential problems and concerns, including preventing dissemination of false information. These meetings will be coordinated by the public health department in the county in strong collaboration with the EGPAF team. Depending on the venue, key stakeholders may include social workers, community health volunteers, local community leaders (chiefs, sub chiefs), members of the county and sub- county health management teams, including those from the public health department, county Coronavirus-19 response manager, county education department, school principals, religious leaders, among others. Ongoing dialogue with these stakeholders will be important to maintain community engagement before and during the study implementation.

A few days before the start of testing campaign, community health volunteers will visit the selected high attendance venues and a poster announcing the community testing activity will be distributed for display in the venue prior to the scheduled testing intervention.

Trained community health volunteers and mobilizers will present to the venue on the pre-agreed day(s) to announce the actual testing day and mobilize the community. Available channels like community, Facebook, and other social media will also be used to mobilize the community. Through church leaders and association of pastors, messages about the testing will be posted on church websites where available. Megaphones and caravans may also be used for community mobilization as deemed appropriate.

Data Collection on the day of testing, individuals accessing the venue will be informed of the SARS-CoV-2 testing taking place and asked if the participants are willing to be tested. An anonymous screening log will be completed for all individuals offered testing, which will include age, sex, whether testing was accepted or not, and any reported reasons for choosing not to test. This will allow capture of a brief description of the population at each venue and documentation of the testing refusal rate.

For those who opt in for testing, the MoH staff will provide routine information on the test procedure before performing the test (see section on testing procedure). During the consenting process, information about the study objectives and procedures will be provided and the client will be able to ask questions. Those who agree will then undergo a 2- to 5-minutes interview. The data obtained from the interview will be recorded in the data collection tool and later entered into the study database.

For individuals tested positive and those negative referred for PCR because of Coronavirus-19 symptoms, the investigators will also collect information on their final PCR result, and the result of their sequencing test after obtaining from them a written informed consent.

PCR/whole genome sequencing (WGS) surveillance:

Kenya Medical Research Institute-Wellcome Trust Research Laboratory in Kilifi is currently the laboratory tasked by the Ministry of Health with SARS-CoV-2 genome sequencing in Kenya. The laboratory operates in compliance with Good Clinical Laboratory Practice (GCLP) standards. For this study, the Coronavirus-19 sequencing sample manifest form (QMS-F238- Annex 5) will be completed with all the required information and sent together with the swabs to Kenya Medical Research Institute-Wellcome Trust Research Laboratory. Laboratory staff will communicate results to the study team using the unique identifiers described above; the study team will update the study database.

Costs will be estimated from a health systems perspective using a micro-costing method, combining top-down and bottom-up approaches to obtain resource use and costs per line item. All project costs will be converted to 2022 U.S. dollars (US$) using the prevailing exchange rate and adjusted to inflation using the U.S. consumer price index if needed.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 2 years
2. Agrees to Undergo testing with SARS-CoV-2-Ag RDT on the day of testing campaign
3. Ability and willingness to provide written consent/assent for participation in an interview following the test

Exclusion Criteria:

* 1. Positive SARS-CoV-2 test done 1 to 14 days before the current testing campaign

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be composed of all persons attending the selected venue where testing is offered on the day of the testing campaign, including all ages > 2 years regardless of presence of coronavirus-19 symptoms. This population will include people from different economic and social backgrounds.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 case detection rate | This will be done in a period of 4 months of study enrolment
  Will determine the proportion of SARS-CoV-2 infections detected per 100 individuals tested) in high volume community venues using SARS-CoV-2 Ag-RDT, overall and disaggregated by venue type.

SECONDARY OUTCOMES:
Proportion testing positive across the cascade | 4 months
  will determine proportion of venue attendees across the SARS-CoV-2 testing cascade
Positive cases by type | 4months
  Proportion of people who test positive with SARS-CoV2 RDT who are symptomatic, are referred for PCR and confirmed with PCR, are referred for home-based isolation or care,
Factors | 4 months
  Factors that are associated with SARS-CoV-2 infection, such as age, venue, exposure history and vaccination status.
SARS-COV-2 variants | 4 months
  SARS-CoV-2 variants among SARS-CoV-2 positive attendees
Costing | 4months
  Costs associated with implementation of SARS-CoV-2 Ag-RDT in community settings.

CONTACTS AND LOCATIONS:
Locations (1):
- Kiambu County, Kiambu, Kenya

IPD SHARING:
Plan to Share IPD: No